CLINICAL TRIAL: NCT04487509
Title: Incidence Study on Acute Coronary Disease With ST Segment Elevation (CAD ST +) in the Emergency Room (InSyCo ST + Study)
Brief Title: Incidence Study on Acute Coronary Disease With ST Segment Elevation
Acronym: InSyCoST+
Status: Completed | Type: Observational
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, PROFESSOR, Hôpital Universitaire Sahloul
Other Study IDs: INSYCO ST+
Record Dates: First submitted 2020-03-28; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Acute Myocardial Infarction; Emergencies; Complication
MeSH Terms: conditions — Emergencies | interventions — Dental Occlusion; Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: THROMBOLYSE — the treatment delivered to the emergency room, in particular the nature of the treatment for obstruction (primary angioplasty or thrombolysis)
  Other Names: OBSTRUCTION; CORONARY ANGIOPLASTY

SUMMARY:
Cardiovascular disease, and in particular ischemic heart disease, is the main cause of morbidity and mortality worldwide today (1). Myocardial infarction (MI) presents the most serious clinical entity through its short-term life threatening involvement.

The many advances in the management of IDM during the acute phase, namely the increasingly frequent and effective use of reperfusion means (angioplasty and thrombolysis) as well as pharmacological progress, in particular, the management of anti-thrombotic treatment has enabled a significant reduction in intra-hospital mortality, in the medium and long term (2). In fact, the mortality rate dropped from 25-30% before the creation of the cardiac intensive care units (ICUS) around the 1960s, to around 16% in the 1980s and reaching 4 to 6% today. In the latest data from the French FAST MI 2015 register (French Registry of Acute ST-Elevation or Non-ST-elevation Myocardial Infarction) mortality was 2.8% in hospital (3) and 5.3% at 6 months (4). Nevertheless, mortality rates diverge from one register to another and are generally higher compared to randomized controlled clinical trials.

In our country, due to the aging of the Tunisian population (currently the oldest population in Africa), as well as the rise in the prevalence of cardiovascular risk factors (5), the incidence of IDM is clearly increasing. However, our local specificities concerning the management of this pathology and the intra-hospital mortality which results from it, remain little described despite the importance of these data in the development of personalized algorithms and the improvement of the quality of this support.

the management of CAD ST + in the public sector poses more and more efficiency problems and moves away from international recommendations in our country, an assessment of our national situation is necessary.

The objectives of the study are, primary, the incidence of new cases that consult the emergency room for CAD ST + and the treatment delivered to the emergency room, in particular the nature of the treatment for obstruction (primary angioplasty or thrombolysis). Secondary, the evaluation of hospital complications and the future of patients on D30 and after one year from the inclusion's day.

DETAILED DESCRIPTION:
Cardiovascular disease, and in particular ischemic heart disease, is the main cause of morbidity and mortality worldwide today (1). Myocardial infarction (MI) presents the most serious clinical entity through its short-term life threatening involvement.

The many advances in the management of IDM during the acute phase, namely the increasingly frequent and effective use of reperfusion means (angioplasty and thrombolysis) as well as pharmacological progress, in particular, the management of anti-thrombotic treatment has enabled a significant reduction in intra-hospital mortality, in the medium and long term (2). In fact, the mortality rate dropped from 25-30% before the creation of the cardiac intensive care units (ICUS) around the 1960s, to around 16% in the 1980s and reaching 4 to 6% today. In the latest data from the French FAST MI 2015 register (French Registry of Acute ST-Elevation or Non-ST-elevation Myocardial Infarction) mortality was 2.8% in hospital (3) and 5.3% at 6 months (4). Nevertheless, mortality rates diverge from one register to another and are generally higher compared to randomized controlled clinical trials.

In our country, due to the aging of the Tunisian population (currently the oldest population in Africa), as well as the rise in the prevalence of cardiovascular risk factors (5), the incidence of IDM is clearly increasing. However, our local specificities concerning the management of this pathology and the intra-hospital mortality which results from it, remain little described despite the importance of these data in the development of personalized algorithms and the improvement of the quality of this support.

the management of CAD ST + in the public sector poses more and more efficiency problems and moves away from international recommendations in our country, an assessment of our national situation is necessary.

The objectives of the study are, primary, the incidence of new cases that consult the emergency room for CAD ST + and the treatment delivered to the emergency room, in particular the nature of the treatment for obstruction (primary angioplasty or thrombolysis). Secondary, the evaluation of hospital complications and the future of patients on D30 and after one year from the inclusion's day.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Acute ST + coronary syndrome, with an ST segment elevation on the ECG at point J in two contiguous leads with the following thresholds: ≥0.1 mv in all leads except V2- V3 where the thresholds will be: ≥ 0.2 mV in men ≥ 40 years old; ≥ 0.25 mV in men.

Exclusion Criteria:

* ST plus equivalents (IVA syndrome, left branch block, etc.),
* CAD without ST segment elevation
* Patients arriving in cardiac arrest and not recovered after resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty four emergency departments are affected in this study for the recruitment of patients. Two months from October 17th to December 17th for the inclusion of patients including public holidays 24 hours 7 days a week plus a month of follow up.
  Data collection Parameters of history (history) Schedules for clinical examinations (triage, ECG) Treatments received in the emergency room Thrombolysis, specifying the schedule and the molecule used Angioplasty, specifying the time and place Complication in the emergency room (death, shock, abortion, rhythm disorder) Transfer and hospital complications Becoming and coming from patients by a phone call Specify previous complications (death, shock, abortion, rhythm disorder) Duration of hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
MORTALITY | one month
  Mortality will be reported.

SECONDARY OUTCOMES:
CORONARY ANGIOPLASTY | one month
  Angioplasty will be reported.
COMPLICATIONS | one month
  Complications will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Boukef Riadh, professor, Principal Investigator — HU Sahloul
Locations (1):
- HU Sahloul, sousse, Tunisia, Sousse, Itinéraire Ceinture Cité Sahloul, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addad F, Mahdhaoui A, Gouider J, Boughzela E, Kamoun S, Boujnah MR, Haouala H, Gamra H, Maatouk F, Ben Khalfallah A, Kachboura S, Baccar H, Ben Halima N, Guesmi A, Sayahi K, Sdiri W, Neji A, Bouakez A, Milouchi S, Battikh K, Jullieres Y, Danchin N, Monsuez JJ, Mulak G, Hagege A, Bataille V, Chettaoui R, Mourali MS; FAST-MI Tunisia investigators. Management of patients with acute ST-elevation myocardial infarction: Results of the FAST-MI Tunisia Registry. PLoS One. 2019 Feb 22;14(2):e0207979. doi: 10.1371/journal.pone.0207979. eCollection 2019. PMID 30794566
- [Background] Trebouet E, Boiffard E, Debierre V, Fradin P. [Analysis of cardiovascular complications occurring during inter-hospital transfers of patients with non-ST elevation myocardial infarction]. Ann Cardiol Angeiol (Paris). 2019 Feb;68(1):13-16. doi: 10.1016/j.ancard.2018.08.019. Epub 2018 Oct 2. French. PMID 30290916